CLINICAL TRIAL: NCT05455970
Title: Effect of Rhythmic Auditory Stimulation on Functional Balance in Children With Cerebral Palsy, A Randomized Control Trial.
Brief Title: Effect of Rhythmic Auditory Stimulation on Balance in Children With Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Apiphan Iamchaimongkol, MD, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ramathibodi
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy, Rhythmic Auditory Stimulation, Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic auditory stimulation (RAS) group (Experimental): Physical therapy including stretching and strengthening exercise and ambulation training with rhythmic auditory stimulation.
  Interventions: Other: Rhythmic auditory stimulation (RAS)
- Conventional group (No Intervention): Conventional physical therapy including stretching exercise, strengthening exercise and ambulation training.

INTERVENTIONS:
Other: Rhythmic auditory stimulation (RAS) — A therapeutic application of pulsed rhythmic or musical stimulation in order to improve gait or movement
  Arms: Rhythmic auditory stimulation (RAS) group

SUMMARY:
To evaluate the effect of Rhythmic Auditory Stimulation (RAS) on balance in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebral palsy at 7-15 years old with Gross motor function classification system 1-3.
* Patients can understand and follow to command.

Exclusion Criteria:

* Patients who received surgery/chemo-denervation injection/injury at spine/pelvic/lower extremities in last 6 months.
* Patients with intrathecal baclofen pump implantation.
* Patients with other signs and/or symptoms of neurological deficit that effect ability to ambulation.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Timed up and go - in children | Change from baseline Timed up and go - in children at after intervention 3 weeks
  The tool to assess functional mobility in pediatric population. This is a timed measure during which the child has to stand up from a chair, walk 3 m, turn around, walk back, and sit down. Higher timed measure mean worse outcome.

SECONDARY OUTCOMES:
Pediatric Balance Scale | Change from baseline Pediatric Balance Scale at after intervention 3 weeks
  A modified version of the Berg Balance Scale from 0-56. That is used to assess functional balance skills in children. Higher scores mean better outcome.
Gross Motor Function Measure | Change from baseline Gross Motor Function Measure at after intervention 3 weeks
  The tool to evaluate gross motor function in children with cerebral palsy. The score from 0-186. Higher scores mean better outcome.
Gait Velocity | Change from baseline Gait Velocity at after intervention 3 weeks
  Gait speed used by 10 meter test recorded in Kilometer per hour. Higher timed measure mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of rhythmic auditory stimulation on gait performance in children with spastic cerebral palsy — https://pubmed.ncbi.nlm.nih.gov/17645385/
- See also: Differential effects of rhythmic auditory stimulation and neurodevelopmental treatment/Bobath on gait patterns in adults with cerebral palsy: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/22308559/
- See also: Changes in gait patterns with rhythmic auditory stimulation in adults with cerebral palsy — https://pubmed.ncbi.nlm.nih.gov/22142756/
- See also: Effects of the Combination of Music Therapy and Physiotherapy in the Improvement of Motor Function in Cerebral Palsy: A Challenge for Research — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8534581/